CLINICAL TRIAL: NCT06987045
Title: Trans and Non-binary Prostate-Specific Antigen Reference Interval Determination Study
Acronym: TransPRIDE
Status: Not yet recruiting | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 336982
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Prostate CA
Keywords: Prostate Cancer; Transwomen; Non-binary; prostate
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 40-49 year olds
- 50-59 year olds
- 60-79 year olds
- 70+ year olds

SUMMARY:
The prostate specific antigen (PSA) blood test can help diagnose prostate problems, including cancer.

The prostate is an organ in the pelvis. It is found in cisgender men, transgender (trans) women and some non-binary people.

Anyone with a prostate can get prostate cancer. The prostate remains after genital (lower) surgery. The hormones and surgeries that trans women and non-binary people might have can lower the PSA. We do not have good data on the normal PSA levels are for this group

TransPRIDE is a research study that will help us find the normal levels of PSA in trans women and non-binary people with prostates.

Researchers will ask 500 trans women and non-binary people with prostates to take part. They will need to be aged 40 or over. They will need to be on hormones or have had lower surgery. They will be called after 6 months to recheck their health. If a person has a high PSA, they may be sent for more tests.

Knowing the normal PSA level for trans women and non-binary people will help doctors to find and treat their prostate cancer more quickly.

ELIGIBILITY:
Inclusion Criteria:

* • Aged >40

  * Transgender or non-binary (identify with a gender other than the one assigned at birth)
  * With a prostate
  * Fulfills at least one of the following 3 criteria with regards to gender-affirming medical care:

    * Taking oestradiol for at least the last 3 months
    * Taking anti-androgens for at least the last 3 months
    * Ever had bilateral orchidectomy
  * Eligible for National Health Service (NHS) treatment

Exclusion Criteria:

* • History of prostate cancer (Prostate cancer) at any time

  * History of prostate surgery at any time
  * History of prostate radiotherapy at any time
  * History of benign prostatic hypertrophy (enlarged prostate) at any time
  * Vaginoplasty within 12 months
  * Orchidectomy or vulvoplasty within three months
  * Sexually Transmitted Infection (STI) within 6 weeks of blood sample
  * Active urinary infection or within 6 weeks of blood sample
  * Prostatitis within 6 weeks of blood sample
  * Urological intervention (e.g. prostate biopsy) within 6 weeks of blood sample
  * Unwilling to give consent
  * Lacking capacity to give consent
  * In the secure estate

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Trans and non-binary people with a prostate (TNBPP) who are taking Gender-Affirming Hormone Therapy (GAHT) and/or have had bilateral orchidectomy.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-10-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is blood PSA concentration. | 6months following end of enrolment
  The 95th percentile will be used to define the upper reference value of PSA values in healthy individuals; this will be estimated separately for each age group (i.e. 40-49, 50-59, 60-79, 70+).

SECONDARY OUTCOMES:
Prostate Cancer | 6months following end of enrolment
  The numbers of participants diagnosed with prostate cancer during the study.

IPD SHARING:
Plan to Share IPD: No